CLINICAL TRIAL: NCT03937362
Title: Accuracy of Detecting Residual Disease After Neoadjuvant Chemoradiotherapy for Esophageal Squamous Cell Carcinoma: the preSINO Trial (Pre-Surgery If Needed for Oesophageal Cancer)
Brief Title: Pre-Surgery If Needed for Oesophageal Cancer
Acronym: preSINO
Status: Completed | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Queen Mary Hospital, Hong Kong (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Zhigang Li, Chief, Shanghai Chest Hospital
Other Study IDs: Chest201902
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; Neoadjuvant chemoradiotherapy; Esophageal cancer; Esophageal squamous cell carcinoma; Active surveillance
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Before neoadjuvant chemoradiotherapy (nCRT), tumor tissues from formalin-fixed paraffin-embedded samples from endoscopy biopsy were collected for whole-exome sequenced for patient-specific somatic variants; then, a personalized panel for circulating tumor DNA (ctDNA) was designed accordingly. Serial peripheral blood samples were collected at 3-5 time points (baseline, CRE-1, CRE-2, 1 month post-surgery, and 3-6 months post-surgery) for ctDNA detection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Clinical Response Evaluation: Patients with operable esophageal squamous cell carcinoma who are planned to undergo neoadjuvant chemoradiotherapy according to the CROSS regimen (intravenous carboplatin AUC 2 mg/mL/min and intravenous paclitaxel 50 mg/m2 on days 1, 8, 15, 22 and 29 with concurrent 41.4 Gy radiotherapy given in 23 fractions of 1.8 Gy on 5 days per week) followed by surgery.
  Patients will undergo a first clinical response evaluation (CRE-1) 4-6 week after completion of nCRT. In patients without histological evidence of residual tumor surgery will be postponed another 6 weeks. A second clinical response evaluation (CRE-2) will be performed 10-12 weeks after completion of nCRT. Immediately after CRE-2 all patients without evidence of distant metastases will undergo esophagectomy.
  Interventions: Diagnostic Test: First clinical response evaluation (CRE-1); Diagnostic Test: Second clinical response evaluation (CRE-2)

INTERVENTIONS:
Diagnostic Test: First clinical response evaluation (CRE-1) — Consisting of: endoscopy with bite-on-bite biopsies
Diagnostic Test: Second clinical response evaluation (CRE-2) — Consisting of: PET-CT, endoscopic bite-on-bite biopsies,EUS with FNA

SUMMARY:
A prospective, multi-centre, diagnostic cohort study investigating the accuracy of positron emission tomography with computed tomography (PET-CT), endoscopic bite-on-bite biopsies and endoscopic ultrasonography (EUS) with fine-needle aspiration (FNA) for detecting residual disease after neoadjuvant chemoradiotherapy in patients with potentially resectable esophageal squamous cell carcinoma (SCC).

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCRT) followed by esophagectomy is a standard treatment for locally-advanced esophageal cancer. After nCRT, high pathologically complete response (pCR) rates are being achieved in patients with esophageal cancer, especially squamous cell carcinoma (SCC). Surgery for esophageal cancer is risky and is associated with reduced quality of life. It is important to know that with an accurate and safe clinical evaluation strategy, some patients might delay surgery or avoid unnecessary surgery and be safely monitored instead. Therefore, an active surveillance strategy has been proposed for patients with clinically complete response (cCR) after nCRT.

The previous European preSANO trial (Lancet Oncol. 2018 Jul;19(7):965-974, PMID: 29861116) showed that the clinical response evaluations (CRE) were sufficiently accurate to detect residual tumor after nCRT in patients with mainly adenocarcinoma, however, its applicability to SCC, which is characterized by extensive lymph node metastasis, remains unknown.

The objective of this study is to assess the accuracy of response evaluations after nCRT based on the preSANO trial, including positron emission tomography with computed tomography (PET-CT), endoscopic bite-on-bite biopsies and endoscopic ultrasonography (EUS) with fine-needle aspiration (FNA) in patients with potentially operable esophageal SCC. Additionally, this study also explores the value of circulating-tumor DNA (ctDNA) in predicting residual disease.

Locally-advanced operable esophageal SCC patients who are planned to undergo nCRT according to the CROSS regimen and are planned to undergo surgery will be recruited from three high-volume Asian centers. Four to six weeks after completion of nCRT, patients will undergo a first clinical response evaluation (CRE-1) consisting of endoscopic bite-on-bite biopsies. In patients without histological evidence of residual tumor (i.e. without positive biopsies), surgery will be postponed another six weeks. A second clinical response evaluation (CRE-2) will be performed 10-12 weeks after completion of nCRT, consisting of PET-CT, endoscopic bite-on-bite biopsies and EUS with FNA. After CRE-2, all patients without evidence of distant metastases will undergo esophagectomy. Primary endpoint is the accuracy of CRE for detecting TRG3-4 or TRG1-2 with ypN+ residual tumor with a prespecified false-negative rate of 19.5%.

Secondary endpoint includes the accuracy of detecting any residual tumor. Exploratory analyses of ctDNA will be performed in patients with available blood samples.

If the current study shows that major residual disease (>10% residual carcinoma at the primary tumor site and any residual nodal disease) can be accurately (i.e. with sensitivity of 80.5%) detected in patients with esophageal SCC, a prospective trial will be conducted comparing active surveillance with standard esophagectomy in patients with a clinically complete response after nCRT (SINO trial).

ELIGIBILITY:
Inclusion criteria are:

1. Histologically confirmed esophageal squamous cell carcinoma;
2. Tumor located in the chest;
3. Clinical stage cT1N1-2M0, cT2-4aN0-2M0, according to the 8th Edition of the AJCC TNM classification for Esophageal Cancer;
4. Age > 20 at the date of informed consent;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of two or less;
6. Considered fit to undergo nCRT followed by surgical resection;
7. Expected survival time more than three months;
8. Written informed consent by the patient.

Exclusion criteria are:

1. Patient with a second primary tumor;
2. Previous major surgery in the chest or upper abdomen;
3. Tumor not 18F-FDG-avid at baseline PET-CT;
4. Suspected positive lymph nodes that cannot be covered by an uninterrupted radiation field that also includes the primary tumor area;
5. Primary (early) lesion already removed by EMR/ESD;
6. Previous history of chemotherapy and/or radiation therapy;
7. Cervical esophageal cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer patients who are planned to undergo nCRT according to the CROSS regimen and who will undergo surgical resection will be recruited from four Asian centres.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of clinical response evaluations for detecting substantial residual locoregional disease | 10-12 weeks after completion of neoadjuvant chemoradiotherapy
  The diagnostic performance in terms of sensitivity and specificity of both CRE-1 and CRE-2 for detecting TRG 3-4 residual tumor (more than 10% residual carcinoma) or TRG 1-2 residual tumor (less than 10% residual carcinoma) with residual nodal disease (ypN+) in the surgical resection specimen.

SECONDARY OUTCOMES:
Accuracy of clinical response evaluations for detecting any residual locoregional disease | 10-12 weeks after completion of neoadjuvant chemoradiotherapy
  The diagnostic performance in terms of sensitivity and specificity of both CRE-1 and CRE-2 for detecting pathologically non-complete response in both the primary tumor and the regional lymph nodes (TRG2-4 or ypN+).

OTHER OUTCOMES:
Accuracy of ctDNA for detecting residual disease after neoadjuvant chemoradiotherapy but prior to surgery | 10-12 weeks after completion of neoadjuvant chemoradiotherapy
  The ctDNA status during CRE-1 and CRE-2 time points will be assessed using a tumor-informed personalized-panel based on next-generation sequencing. The diagnostic performance in terms of sensitivity and false-nageative of the combination of biopsy and ctDNA for detecting residual tumor in the surgical resection specimen
Prognostic value of ctDNA for predicting disease-free survival | 1 year after completion of neoadjuvant chemoradiotherapy and surgery
  The postoperative ctDNA status will be assessed using a tumor-informed personalized-panel based on next-generation sequencing. Patients will be stratified according to their ctDNA status. Disease-free survival is defined as the time from the completion of treatment to recurrence or death from any cause. Survival prognostic analyses will adjust for clinical factors and TNM staging using Cox regression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Li, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (4):
- Shanghai Chest Hospital, Shanghai, China
- Queen Mary Hospital, Hong Kong, Hong Kong
- Erasmus MC Cancer Institute, Rotterdam, Netherlands
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang X, Eyck BM, Yang Y, Liu J, Chao YK, Hou MM, Hung TM, Pang Q, Yu ZT, Jiang H, Law S, Wong I, Lam KO, van der Wilk BJ, van der Gaast A, Spaander MCW, Valkema R, Lagarde SM, Wijnhoven BPL, van Lanschot JJB, Li Z. Accuracy of detecting residual disease after neoadjuvant chemoradiotherapy for esophageal squamous cell carcinoma (preSINO trial): a prospective multicenter diagnostic cohort study. BMC Cancer. 2020 Mar 6;20(1):194. doi: 10.1186/s12885-020-6669-y. PMID 32143580
- [Derived] Liu Z, Wang G, Yang Y, Su Y, Zhang H, Liu J, Cui P, Fan X, Yang J, Zhang Z, Gao X, Chao Y, Mostert B, van Lanschot JJB, Wijnhoven BPL, Law S, Li C, Cai S, Li Z. ctDNA detects residual disease after neoadjuvant chemoradiotherapy and guides adjuvant therapy in esophageal squamous cell carcinoma. Cell Rep Med. 2025 Sep 16;6(9):102334. doi: 10.1016/j.xcrm.2025.102334. Epub 2025 Sep 5. PMID 40914168